CLINICAL TRIAL: NCT07259330
Title: A Phase 1, Single-Sequence, Two-Period Crossover, Open-Label Study to Determine the Potential Induction Effect of Multiple 100 mg BID Oral Doses of Nirogacestat on a Cocktail of CYP Probe Substrates CYP2B6 (Bupropion), CYP2C8 (Repaglinide), CYP2C9 (Flurbiprofen), CYP2C19 (Omeprazole), and CYP3A4 (Midazolam) in Healthy Males
Brief Title: To Determine the Effect of CYP Induction Following Administration of Nirogacestat in Healthy Adult Male Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NIR-DT-106; 2025-521402-18-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-19; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Healthy
MeSH Terms: interventions — nirogacestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nirogacestat (Active Comparator): Nirogacestat 100 mg BID will be administered orally from Day 1 through Day 17
  Interventions: Drug: Nirogacestat
- Nirogacestat and CYP cocktail (Experimental): Nirogacestat 100 mg BID will be administered orally from Day 1 through Day 17 and an oral dose of CYP cocktail (CYP2B6 [bupropion 20 mg], CYP2C8 [repaglinide 0.05 mg], CYP2C9 [flurbiprofen 10 mg], CYP2C19 [omeprazole 10 mg], and CYP3A4 [midazolam 1 mg]) will be administered on Day -3, and again on Day 15.
  Interventions: Drug: Nirogacestat and Cocktail of CYP Specific Probe Substrates

INTERVENTIONS:
Drug: Nirogacestat — 100 mg tablet Day 1 through Day 17
  Arms: Nirogacestat
Drug: Nirogacestat and Cocktail of CYP Specific Probe Substrates — Drug: Nirogacestat 100 mg tablet Day 1 through Day 17 and Drug: Cocktail of CYP Specific Probe Substrates administered Day 15.
  Arms: Nirogacestat and CYP cocktail

SUMMARY:
This study will evaluate the effects of nirogacestat 100 mg twice daily (BID) on the pharmacokinetics (PK) of a cytochrome P450 (CYP) cocktail.

DETAILED DESCRIPTION:
This is a single-center, single-sequence crossover study to assess the potential induction effects of nirogacestat on the PK of probe substrates for CYPs (CYP2B6, CYP2C8, CYP2C9, CYP2C19, and CYP3A4) in healthy adult men.

There will be a Screening Period of up to 33 days prior to Day -4. Eligible participants will be enrolled in the study and will complete a 3-day Lead-In Period, followed by an 18-day Treatment Period. A follow-up (FU) telephone call will be performed 26 to 28 days after the last dose of study treatment (Day 43 [+2]).

During Screening, participants will sign the informed consent form prior to any study procedures being performed. Participants must satisfy all the inclusion and exclusion criteria to be eligible for study participation. Participants will be admitted to the clinical research unit (CRU) on Day -4 for check-in procedures and eligibility confirmation.

Once eligibility is confirmed, participants will receive a CYP cocktail (CYP2B6 [bupropion], CYP2C8 [repaglinide], CYP2C9 [flurbiprofen], CYP2C19 [omeprazole], and CYP3A4 [midazolam]) on the morning of Day -3, following an overnight fast of at least 10 hours. The CYP cocktail will be administered orally.

Beginning on Day 1 through Day 17, participants will be administered 100 mg nirogacestat orally BID. On Day 15, following an overnight fast of at least 10 hours, participants will also receive a single oral dose of the CYP cocktail in the morning immediately following the oral dose of nirogacestat. On all other days, nirogacestat can be administered with or without food. Study treatment will be administered orally.

Assessments for safety along with serial samples of blood will be collected throughout the Lead-In and Treatment Period.

Participants will remain domiciled at the CRU until all safety evaluations are completed on Day 18.

Participants will complete a FU telephone visit on Day 43 (+2 days) for review of AEs/serious AEs and concomitant medications. Additional safety evaluations may be scheduled at the discretion of the investigator prior to the FU telephone visit.

ELIGIBILITY:
Inclusion Criteria:

1. Participant understands the study procedures, is willing to comply with all study requirements and restrictions and agrees to participate in the study by providing written informed consent prior to any study-related procedures being performed.
2. Participant is a male between 18 and 55 years of age (inclusive) at the time of informed consent.
3. Participant has a body mass index (BMI) ≥18 kg/m2 and ≤32 kg/m2 (inclusive) at Screening and Day -4, and a total body weight >50 kg.
4. Participant is considered to be medically healthy, as determined by a responsible and experienced investigator, based on a clinical evaluation (including medical history, physical examination, clinical laboratory tests, vital sign measurements, and a 12-lead electrocardiogram [ECG] and the results of clinical chemistry coagulation and urinalysis carried out at Screening and Day -4.
5. Participant has alanine aminotransferase, aspartate aminotransferase, and total bilirubin levels less than 1.5×the upper limit of normal at Screening and at Day -4.
6. Participant has a renal function (creatinine clearance ≥90 mL/min), as evidenced by normal estimated glomerular filtration rate measured by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation at Screening and at Day -4.
7. Participants that agree to the following during the Treatment Period, and for at least 7 days after the last dose of study treatment:

   1. Refrain from donating or preserving sperm; PLUS either
   2. Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent.

   OR c. Must agree to use a male condom when having sexual intercourse with women of childbearing potential (WOCBP). An additional form of contraception must also be used by the female partner if she is of childbearing potential.
8. Has sufficiently good venous access in at least 1 arm to confidently enable serial blood sampling.

Exclusion Criteria:

* 1. Participant has a history or presence of oncologic, cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, ocular, endocrine, immunologic, dermatologic, musculoskeletal, neurologic, psychiatric, or other disease or condition or the laboratory test abnormality that, in the investigator's judgment, poses a significant risk to the safety of the participant or the achievement of study objectives.

  2. Participant has a history or presence of any condition possibly affecting drug absorption (e.g., gastrectomy).

  3. Participant has a medical history or abnormal findings at Screening or Day -4 that the investigator judges may put at risk achieving the objectives of the study or protecting the safety of the participant.

  4. Participant has an acute illness with symptoms or treatment that has started or persisted within 14 days prior to study treatment administration, unless mild in severity, and enrollment is approved by both investigator and sponsor's medical monitor.

  5. Participant has tested positive for hepatitis B virus, hepatitis C virus, or HIV, or has a clinically significant infection.

  6. Participant has blood pressure (BP) that is ≥140 mmHg systolic or ≥90 mmHg diastolic following at least 5 minutes of supine rest at Screening or Day -4. Additionally, BP that is <90 mmHg systolic or <45 mmHg diastolic following at least 5 minutes of a supine rest at Screening or Day -4.

  7. Participant has heart rate (HR) that is <40 bpm or >100 bpm after resting in a supine position for 5 minutes at Screening or Day -4.

  8. Participant has averaged QT interval corrected using Fridericia's formula results from valid triplicate ECGs >450 msec at Screening or Day -4.

  9. Participant has family history of long QT syndrome, or of unexplained sudden death or drowning in a first-degree relative under age 50.

  10. Participant has an ECG waveform abnormality that interferes with QT/QTc interval measurement or interpretation. A participant with mild sinus arrhythmia or sparse isolated premature ventricular contractions is eligible at the investigator's discretion.

  11. Participant has a positive serum alcohol test or other drug screen test at Screening and/or Day -4.

  12. Participant has received any vaccine within 14 days prior to the first dose of study treatment administration on Day -3.

  13. Participant has received any CYP3A4 inhibitors or inducers within 21 days or 5 half-lives (whichever is longer) prior to Day -3.

  14. Participant has had concurrent use of, or has used any long-acting gastric acid reducing agents, including histamine-2 receptor antagonists and proton pump inhibitors, including over-the-counter agents, in the last 21 days prior to Day -3.

  15. Participant has received any prescription or nonprescription drugs (including vitamins and dietary or herbal supplements) within 3 weeks or 5 half-lives, if known (whichever is longer), prior to study treatment administration on Day -3, unless in the opinion of the investigator and sponsor that the medication will not interfere with the study.

  16. Participant has received an investigational product within 30 days or 5 times the half-lives, if known, of any drug used in the prior study (whichever is longer), or exposure to >4 new investigational agents within 12 months prior to study treatment administration on Day -3.

  17. Participant has a known hypersensitivity or intolerance to any of the study treatments, or excipients thereof, or a history of drug or other allergy that, in the opinion of the investigator or sponsor medical monitor, contraindicates their participation.

  18. Participant has a history of excessive intake of alcohol, defined as an average an average weekly intake of >21 units (1 unit is equivalent to 1 can or bottle [250 mL] of beer, or 1 measure [35 mL] of spirits, or 1 glass [100 mL] of wine) in the last 6 months prior to Screening.

  19. Participant has a history of illicit drug abuse within the past 2 years prior to Screening.

  20. Participant has consumed red wine or any fruit juices (including, but not limited to, grapefruit, grapefruit juice, pomelos, exotic citrus fruits, or grapefruit hybrids) within 72 hours of Day -4.

  21. Participant has used caffeine or other xanthine containing products (e.g., coffee, black tea, green tea, colas, cacao, guarana, guayusa, yerba mate) within 48 hours of Screening and Day -4.

  22. Participant regularly consumes excessive amounts (defined as >5 cups per day) of caffeine, xanthine-containing products, or energy drinks, as judged by the investigator.

  23. Participant has used tobacco- or nicotine-containing products within 2 months prior to Screening.

  24. Participant has donated blood or had a loss of >450 mL of blood within 60 days, or donation of plasma within 7 days prior to CRU admission on Day-4.

  25. Participant has received blood products within the 60 days prior to Screening.

  26. Participant is unwilling to avoid strenuous or unaccustomed activity, sunbathing, or contact sports within 96 hours prior to admission to the CRU and until discharge from the CRU.

  27. Participant is deemed unsuitable for this study in the opinion of the investigator for any additional reason, condition, or prior therapy.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Plasma area under the concentration-time curve from dosing extrapolated to infinity (AUCinf) and maximum observed plasma concentration (Cmax) for the CYP cocktail probes alone, and coadministered with nirogacestat. | CYP cocktail - Day -3 and Day 15 at predose (-60 minutes) and at 0.5, 1, 2, 3, 4, 6, 8, (10% nominal), 12, 24, 48, and 72 hours and nirogacestat Days 1 through 17 predose trough samples should be obtained within 1 hour of the nominal time from dosing.
  Area under the concentration-time curve from dosing extrapolated to infinity. AUCinf = (AUClast + Clast/Kel) where Clast is the plasma concentration at the last quantifiable timepoint estimated from the log-linear regression analysis and Kel is the terminal elimination phase rate constant estimated by linear regression based on observations justified to describe the terminal phase on the log-linear concentration-time profile.
Maximum Observed Plasma Concentration (Cmax) of the CYP cocktail probes alone, and coadministered with nirogacestat. | CYP cocktail - Day -3 and Day 15 at predose (-60 minutes) and at 0.5, 1, 2, 3, 4, 6, 8, (10% nominal), 12, 24, 48, and 72 hours and nirogacestat Days 1 through 17 predose trough samples should be obtained within 1 hour of the nominal time from dosing.
  Maximum observed plasma concentration. Observed directly from the data.

SECONDARY OUTCOMES:
Plasma AUClast for the CYP cocktail probes alone and coadministered with nirogacestat. | CYP cocktail - Day -3 and Day 15 at predose (-60 minutes) and at 0.5, 1, 2, 3, 4, 6, 8, (10% nominal), 12, 24, 48, and 72 hours and nirogacestat Days 1 through 17 predose trough samples should be obtained within 1 hour of the nominal time from dosing.
  Area under the concentration-time curve from dosing to time of the last quantifiable concentration. Linear-log trapezoidal method.
Plasma time of maximum observed concentration (Tmax) for the CYP cocktail probes alone and coadministered with nirogacestat. | CYP cocktail - Day -3 and Day 15 at predose (-60 minutes) and at 0.5, 1, 2, 3, 4, 6, 8, (10% nominal), 12, 24, 48, and 72 hours and nirogacestat Days 1 through 17 predose trough samples should be obtained within 1 hour of the nominal time from dosing.
  Time of maximum observed concentration. Observed directly from the data as the time of first occurrence of Cmax
Plasma apparent terminal elimination half-life (t1/2) for the CYP cocktail probes alone and coadministered with nirogacestat. | CYP cocktail - Day -3 and Day 15 at predose (-60 minutes) and at 0.5, 1, 2, 3, 4, 6, 8, (10% nominal), 12, 24, 48, and 72 hours and nirogacestat Days 1 through 17 predose trough samples should be obtained within 1 hour of the nominal time from dosing.
  Apparent terminal elimination half-life calculated as ln(2)/Kel.
Plasma apparent oral clearance (CL/F) for the CYP cocktail probes alone and coadministered with nirogacestat. | CYP cocktail - Day -3 and Day 15 at predose (-60 minutes) and at 0.5, 1, 2, 3, 4, 6, 8, (10% nominal), 12, 24, 48, and 72 hours and nirogacestat Days 1 through 17 predose trough samples should be obtained within 1 hour of the nominal time from dosing.
  Apparent oral clearance. Calculated as Dose/AUCinf
Plasma apparent oral volume of distribution (Vd/F) for the CYP cocktail probes alone and coadministered with nirogacestat. | CYP cocktail - Day -3 and Day 15 at predose (-60 minutes) and at 0.5, 1, 2, 3, 4, 6, 8, (10% nominal), 12, 24, 48, and 72 hours and nirogacestat Days 1 through 17 predose trough samples should be obtained within 1 hour of the nominal time from dosing.
  Apparent oral volume of distribution. Calculated as Dose/(AUCinf × Kel).
Plasma AUClast of respective probe substrate metabolites alone and coadministered with nirogacestat and the metabolite(s) to parent molar ratio for AUClast (MRAUClast), AUCinf (MRAUCinf), and Cmax (MRCmax) (as data permit). | CYP cocktail - Day -3 and Day 15 at predose (-60 minutes) and at 0.5, 1, 2, 3, 4, 6, 8, (10% nominal), 12, 24, 48, and 72 hours and nirogacestat Days 1 through 17 predose trough samples should be obtained within 1 hour of the nominal time from dosing.
  Area under the concentration-time curve from dosing to time of the last quantifiable concentration. Linear-log trapezoidal method.
Plasma Cmax of respective probe substrate metabolites alone and coadministered with nirogacestat and the metabolite(s) to parent molar ratio for AUClast (MRAUClast), AUCinf (MRAUCinf), and Cmax (MRCmax) (as data permit). | CYP cocktail - Day -3 and Day 15 at predose (-60 minutes) and at 0.5, 1, 2, 3, 4, 6, 8, (10% nominal), 12, 24, 48, and 72 hours and nirogacestat Days 1 through 17 predose trough samples should be obtained within 1 hour of the nominal time from dosing.
  Maximum observed plasma concentration. Observed directly from the data.
Plasma Tmax of respective probe substrate metabolites alone and coadministered with nirogacestat and the metabolite(s) to parent molar ratio for AUClast (MRAUClast), AUCinf (MRAUCinf), and Cmax (MRCmax) (as data permit). | CYP cocktail - Day -3 and Day 15 at predose (-60 minutes) and at 0.5, 1, 2, 3, 4, 6, 8, (10% nominal), 12, 24, 48, and 72 hours and nirogacestat Days 1 through 17 predose trough samples should be obtained within 1 hour of the nominal time from dosing.
  Time of maximum observed concentration. Observed directly from the data as the time of first occurrence of Cmax.
Serum nirogacestat, trough concentration (Ctrough). | Days 1 through 17 predose trough samples should be obtained within 1 hour of the nominal time from dosing.
  Pre-dose concentration. Observed directly from the data.
Number of participants with Adverse Events | Baseline (Day -4) through the Follow-up Phone Call (Day 43)
  An adverse event (AE) was defined as any untoward medical occurrence in a participant. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a study intervention. A serious adverse event (SAE) was any untoward medical occurrence that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important.
Number of Participants With Clinically Meaningful Change From Baseline in Laboratory Values | Baseline (Day -4) through Day 18
  Number of participants with clinically significant change from baseline in laboratory parameters were reported. Clinical Significance was decided by the investigator. Laboratory investigation included hematology, biochemistry, urinalysis, and coagulation.
Number of Participants With Clinically Meaningful Change From Baseline in Vital Signs | Baseline (Day -4) through Day 18
  Number of participants with clinically significant change from baseline in vital signs. Clinical Significance was decided by the investigator. Vital signs included oral body temperature, systolic blood pressure, diastolic blood pressure, and pulse rate.
Number of Participants With Clinically Meaningful Change From Baseline in Electrocardiogram (ECG) | Baseline (Day -4) through Day 18
  Number of participants with clinically significant change from baseline in ECG parameters were reported. Clinical Significance was decided by the investigator. The 12-lead ECGs were recorded after the participants have rested for at least 5 minutes in supine position. The parameters included heart rate (HR), Respiratory Rate, Pulse Rate, QRS, QT, QTcB and QTcF
Number of Participants With Clinically Meaningful Change From Baseline in Physical Exams | Baseline (Day -4) through Day 18
  A comprehensive physical examination will include, at a minimum, assessments of the cardiovascular, respiratory, gastrointestinal, and neurologic systems. Height and weight will also be measured and recorded. A symptom-directed physical examination will include, at a minimum, assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen).

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen van de Wetering, MD, Principal Investigator — ICON plc
Locations (1):
- ICON Martini Groningen CRU, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No